CLINICAL TRIAL: NCT04399694
Title: Identification and Characterization of Novel Coding, Splicing and Non-Coding Variants That Contribute to Genetic Disorders
Brief Title: Identification and Characterization of Novel Non-Coding Variants That Contribute to Genetic Disorders
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00090878
Record Dates: First submitted 2020-05-15; First posted 2020-05-22 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Genetic Disease; Inborn Errors of Metabolism; Glycogen Storage Disease; Lysosomal Storage Diseases; Storage Disease
MeSH Terms: conditions — Genetic Diseases, Inborn; Metabolism, Inborn Errors; Glycogen Storage Disease; Lysosomal Storage Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples with DNA and/or RNA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this study is to identify and characterize novel non-coding and splicing variants that may contribute to genetic disorders. We will particularly focus on patients with a diagnosed genetic disorder that has inconclusive genetic findings.

DETAILED DESCRIPTION:
To perform this study, we will use patient DNA and RNA that is isolated from blood samples. DNA will be sequenced (targeted capture and/or whole genome DNA sequencing (WGS)) to identify any non-coding single nucleotide variants (SNVs), smaller insertions/deletions (indels), or larger structural variants (SVs). RNA will be sequenced (RNA-seq) to identify genes that are expressed in a differential and/or allele-specific manner, which may indicate a functional non-coding or splicing variant. We will test the function of non-coding variants using high-throughput reporter assays and CRISPR based methodologies.

ELIGIBILITY:
Inclusion criteria:

Subjects will have one or more of the following:

* Patients (probands) diagnosed with a genetic disease
* Patients (probands) with inconclusive genetic results
* Patients (probands) that have identical coding and/or splicing variants, but display highly diverse phenotypes
* Unaffected family members of probands

Exclusion Criteria: There are no exclusion criteria for this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with diagnosed genetic disease and inconclusive genetic results and their unaffected family members
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2024-04-11 (Actual); Study Completion 2024-04-11 (Actual)

PRIMARY OUTCOMES:
Number of missing pathogenic protein coding variants | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Priya Kishnani, MD, Principal Investigator — Duke; Greg Crawford, PhD, Principal Investigator — Duke
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be submitted to dbGaP, casual variants to ClinVar, aggregate rare phenotype and variant data to Geno2MP and other databases, candidate genes via a public list and linked to a node of the MatchMaker Exchange (MyGene2).
Supporting Information: CSR
Time Frame: Data will be available 7-12 months after results are generated and will be available forever.